CLINICAL TRIAL: NCT03158961
Title: A Prospective Evaluation of the Feasibility and Safety of the Transoral Endoscopic Thyroidectomy Vestibular Approach (TOETVA) as a Treatment for Benign Thyroid Nodules
Brief Title: The Feasibility and Safety of the TOETVA for Benign Thyroid Nodules
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Dr. Lang Hung Hin, Brian, Clinical Associate Professor, The University of Hong Kong
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UW 17-144
Record Dates: First submitted 2017-05-15; First posted 2017-05-18 (Actual); Last update posted 2021-04-28 (Actual); Status verified 2021-04

CONDITIONS: Thyroid Diseases
Keywords: Thyroid; Thyroidectomy; Transoral; Endoscopic; Surgery
MeSH Terms: conditions — Thyroid Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TOETVA (Experimental): a new approach in surgery which can treat the thyroid disease
  Interventions: Procedure: Transoral endoscopic thyroidectomy vestibular approach

INTERVENTIONS:
Procedure: Transoral endoscopic thyroidectomy vestibular approach — TOVETA is a new approach in surgery of thyroidectomy no longer open on the neck

SUMMARY:
Thyroid surgery has been developed as a new technique for zero scar in surgery by applying transoral endoscopic thyroidectomy with sublingual approach. The new technique is locating the surgery which pierced through floor of mouth, cause severe tissue damage, high complication, and conversion rates to open surgery and surgical difficulties due to limitation of movement. Nevertheless, each report is still including small number of patients. Recently, the transoral endoscopic thyroidectomy vestibular approach (TOETVA) has been proven feasible and safe in several overseas centers. Moreover, a successful TOETVA case was reported in local media in the late last year. Hence, this study is for evaluating the feasibility and safety of the TOETVA prospectively at a tertiary referral center in Hong Kong.

The following are the procedure of the study:

1. Recruit patients from the clinic.
2. Patients will receive treatment within 3 months
3. Patients will have different assessments like Ultrasonography assessment, Fine needle biopsy, Direct laryngoscopy, and Cosmectic scoring in Pre-operation, post-operation 2 week, post 1 month, post 3 month, post 6 month and post 12 month.
4. Patients will be monitoring by the same team after the study.

ELIGIBILITY:
Inclusion Criteria:

* have a cyst, nodule or a goiter which has been shown to be benign on fine needle aspiration cytology,
* need to undergo a unilateral thyroid resection,
* have a nodule size no larger than 4cm in largest diameter,
* willing to undergo this new approach rather than the traditional open approach.

Exclusion Criteria:

* unfit for surgery,
* has had previous surgery or radiation at the neck,
* unable to tolerate a general anesthesia,
* wearing dental braces,
* absence of vocal cord mobility at laryngoscopy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2017-07-01 (Actual); Primary Completion 2019-05-31 (Actual); Study Completion 2019-07-31 (Actual)

PRIMARY OUTCOMES:
The complication rate after TOETVA in 12 months | 12 months
  To record any complication of surgery in every post-operation visit after 12 months. The record will be used for the calculation of complication rate.

SECONDARY OUTCOMES:
The open conversion rate of TOETVA | 12 months
  To record any cases which need to apply open surgery necessary during the procedure of TOETVA
The wound infection rate after TOETVA | 12 months
  To record the situation of wound infection after surgery
The hematoma rate after TOETVA | 12 months
  To record the situation of hematoma after surgery
The vocal cord palsy rate after TOETVA | 12 months
  To calculate the vocal cord situation after surgery within 12 months
The hypoparathyroidism rate after TOETVA | 12 months
  To record the thyroid function from blood test in 12 months after surgery and calculate the rate of hypo-parathyroid function
The pain score of patient after TOETVA | 12 months
  The pain scoring with 0-10 to assess the pain level of having TOETVA
The satisfaction of patients after having TOETVA in 12 months | 12 months
  The satisfaction in 0-10 scoring after the surgery

CONTACTS AND LOCATIONS:
Overall Officials: Hung Hin, Brian Lang, MBBS(Hons), Principal Investigator — The University of Hong Kong
Locations (1):
- Queen Mary Hospital, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hegedus L, Bonnema SJ, Bennedbaek FN. Management of simple nodular goiter: current status and future perspectives. Endocr Rev. 2003 Feb;24(1):102-32. doi: 10.1210/er.2002-0016. PMID 12588812
- [Background] Erdogan MF, Gursoy A, Erdogan G. Natural course of benign thyroid nodules in a moderately iodine-deficient area. Clin Endocrinol (Oxf). 2006 Dec;65(6):767-71. doi: 10.1111/j.1365-2265.2006.02664.x. PMID 17121528
- [Background] Bergenfelz A, Jansson S, Kristoffersson A, Martensson H, Reihner E, Wallin G, Lausen I. Complications to thyroid surgery: results as reported in a database from a multicenter audit comprising 3,660 patients. Langenbecks Arch Surg. 2008 Sep;393(5):667-73. doi: 10.1007/s00423-008-0366-7. Epub 2008 Jul 17. PMID 18633639
- [Background] Lang BH. Minimally invasive thyroid and parathyroid operations: surgical techniques and pearls. Adv Surg. 2010;44:185-98. doi: 10.1016/j.yasu.2010.05.012. PMID 20919522
- [Background] Rattner D, Kalloo A; ASGE/SAGES Working Group. ASGE/SAGES Working Group on Natural Orifice Translumenal Endoscopic Surgery. October 2005. Surg Endosc. 2006 Feb;20(2):329-33. doi: 10.1007/s00464-005-3006-0. No abstract available. PMID 16402290
- [Background] Clark MP, Qayed ES, Kooby DA, Maithel SK, Willingham FF. Natural orifice translumenal endoscopic surgery in humans: a review. Minim Invasive Surg. 2012;2012:189296. doi: 10.1155/2012/189296. Epub 2012 Jun 6. PMID 22720153
- [Background] Witzel K, von Rahden BH, Kaminski C, Stein HJ. Transoral access for endoscopic thyroid resection. Surg Endosc. 2008 Aug;22(8):1871-5. doi: 10.1007/s00464-007-9734-6. Epub 2007 Dec 28. PMID 18163167
- [Background] Benhidjeb T, Wilhelm T, Harlaar J, Kleinrensink GJ, Schneider TA, Stark M. Natural orifice surgery on thyroid gland: totally transoral video-assisted thyroidectomy (TOVAT): report of first experimental results of a new surgical method. Surg Endosc. 2009 May;23(5):1119-20. doi: 10.1007/s00464-009-0347-0. Epub 2009 Mar 5. PMID 19263151
- [Background] Wilhelm T, Metzig A. Video. Endoscopic minimally invasive thyroidectomy: first clinical experience. Surg Endosc. 2010 Jul;24(7):1757-8. doi: 10.1007/s00464-009-0820-9. Epub 2009 Dec 25. PMID 20035350
- [Background] Wilhelm T, Metzig A. Endoscopic minimally invasive thyroidectomy (eMIT): a prospective proof-of-concept study in humans. World J Surg. 2011 Mar;35(3):543-51. doi: 10.1007/s00268-010-0846-0. PMID 21088839
- [Background] Anuwong A. Transoral Endoscopic Thyroidectomy Vestibular Approach: A Series of the First 60 Human Cases. World J Surg. 2016 Mar;40(3):491-7. doi: 10.1007/s00268-015-3320-1. PMID 26546193
- [Background] Inabnet WB 3rd, Suh H, Fernandez-Ranvier G. Transoral endoscopic thyroidectomy vestibular approach with intraoperative nerve monitoring. Surg Endosc. 2017 Jul;31(7):3030. doi: 10.1007/s00464-016-5322-y. Epub 2016 Nov 10. PMID 27834022
- [Background] Udelsman R, Anuwong A, Oprea AD, Rhodes A, Prasad M, Sansone M, Brooks C, Donovan PI, Jannitto C, Carling T. Trans-oral Vestibular Endocrine Surgery: A New Technique in the United States. Ann Surg. 2016 Dec;264(6):e13-e16. doi: 10.1097/SLA.0000000000002001. No abstract available. PMID 27649533